CLINICAL TRIAL: NCT03753945
Title: Spine MRI in Patients With Deep Brain Stimulation (DBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-6176
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease; Dystonia; Depression; Spinal Stenosis; Spinal Diseases
Keywords: deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Dystonia; Depression; Spinal Stenosis; Spinal Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study that will enroll patients who have already undergone DBS electrode placement for a variety of disorders including, but not limited to Parkinson's disease, essential tremor, dystonia, depression, epilepsy, neuropathic pain and Alzheimer's disease. This eligible patient population is broad but unified by the fact that they have undergone DBS to treat specific circuit dysfunctions. Patients with internalized leads and IPG may be included. Patients will undergo routine clinical MRI sequences used for the spine (structural in axial and sagittal planes). The choice of imaging the cervical, thoracic or lumbar will depend on the requisition from the treating physician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DBS electrode placement (Experimental): Participants in this study will be patients who have already undergone surgery for implantation of DBS electrodes.
  Patients who have already undergone surgery for implantation of DBS electrodes and patients for whom the treating physicians recommends (based on clinical grounds) a spine MRI (cervical, thoracic or lumbar) shall be recruited for the study.This eligible patient population is broad but unified by the fact that they have undergone DBS to treat specific circuit dysfunctions. Patients with internalized leads and IPG may be included. Patients will undergo routine clinical MRI sequences used for the spine (structural in axial and sagittal planes). The choice of imaging the cervical, thoracic or lumbar will depend on the requisition from the treating physician.
  Interventions: Diagnostic Test: MRI of the spine

INTERVENTIONS:
Diagnostic Test: MRI of the spine — Perform a clinically indicated MRI of the spine in DBS patients

SUMMARY:
Magnetic resonance imaging (MRI) of patients implanted with deep brain stimulation (DBS) is under strict safety guidelines. Depending on the body part being imaged, the safety may vary.

Many DBS patients will need a spine MRI based on their clinical symptoms. However, the vendor safety guidelines are limiting in terms of possible MR pulse sequences. Based on phantom safety data, we designed a set of MR pulse sequences deemed as safe as possible and the protocol allows acquisition of diagnostic quality MRI images.

DETAILED DESCRIPTION:
The patients who clinically require a spine MRI will undergo a spine MRI with our designed protocols to obtain diagnostic quality images. Furthermore, a limited brain MRI will be done before and after to ensure no peri-electrode tissue changes.

ELIGIBILITY:
Inclusion criteria

* Age between 18 and 85 years of age
* Participants must have undergone implantation of DBS electrodes.
* Participants must be able to understand the purpose of this research and must sign the informed consent form.
* Participants must understand that the role of this research is demonstrate the safety of spine MRI in patients with DBS.

Exclusion criteria

* Participants who have serious cognitive or psychological impairments and cannot give informed consent.
* Participants who are unable to effectively or efficiently communicate, for example patients suffering from speech deficits (dysarthria, aphasia) or are non-English speaking.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of MRI-related Adverse Events [Safety] | Immediately after the MRI
  Assess for adverse events as seen on clinical examination

SECONDARY OUTCOMES:
Assessment of Peri-electrode Tissue Changes (MRI) | Immediately after the MRI
  Assess for peri-electrode tissue changes as seen on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Boutet A, Elias GJB, Gramer R, Neudorfer C, Germann J, Naheed A, Bennett N, Li B, Gwun D, Chow CT, Maciel R, Valencia A, Fasano A, Munhoz RP, Foltz W, Mikulis D, Hancu I, Kalia SK, Hodaie M, Kucharczyk W, Lozano AM. Safety assessment of spine MRI in deep brain stimulation patients. J Neurosurg Spine. 2020 Feb 14;32(6):973-983. doi: 10.3171/2019.12.SPINE191241. Print 2020 Jun 1. PMID 32059193